CLINICAL TRIAL: NCT04294485
Title: Physical Therapy Intervention in Hospitalized Pleural Effusion Patients
Brief Title: Physical Therapy Intervention in Pleural Effusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0085UG
Record Dates: First submitted 2019-11-12; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Pleural Effusion
Keywords: Physical therapy; Pleural effusion
MeSH Terms: conditions — Pleural Effusion | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Physical therapy intervention Efficacy of electrostimulation intervention combined with lower limbs exercise.
  Interventions: Behavioral: Physical therapy
- Control group (No Intervention): Participants will no receive physical therapy intervention

INTERVENTIONS:
Behavioral: Physical therapy — Electrostimulation combined with exercise
  Arms: Experimental group

SUMMARY:
To know the effects of a physical therapy intervention in patients hospitalized with pleural effusion. The investigators will study the effects of the intervention in hospital stay, health status, psychologica distress and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were pleural effusion patients hospitalized.

Exclusion Criteria:

* Inability to provide informed consent.
* Presence of psychiatric or cognitive disorders.
* Progressive neurological disorders, organ failure, or inability to cooperate.
* Patients who had experienced another pleural effusion in the previous month.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-28 (Estimated); Primary Completion 2020-06-12 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
EuroQol-5 Dimensions visual analogue scale score | Baseline
  European Quality of Life questionnaire consists of the EQ-5D visual analog scale. The visual analog scale has a rating scale of 0-100 (0 worst possible health, and 100 best possible health).
EuroQol-5 Dimensions visual analogue scale score | Up to 7 days
  European Quality of Life questionnaire consists of the EQ-5D visual analog scale. The visual analog scale has a rating scale of 0-100 (0 worst possible health, and 100 best possible health).
EuroQol-5 Dimensions visual analogue scale score | Up to 3 months
  European Quality of Life questionnaire consists of the EQ-5D visual analog scale. The visual analog scale has a rating scale of 0-100 (0 worst possible health, and 100 best possible health).
EuroQol-5 Dimensions index score | Baseline
  European Quality of Life questionnaire consists of the EQ-5D index. The questionnaire has 5 domains: mobility, self-care, usual activity, pain, and anxiety-depression. For each item, the subject selects one of 3 descriptive health states (from good to poor).
EuroQol-5 Dimensions index score | Up to 7 days
  European Quality of Life questionnaire consists of the EQ-5D index. The questionnaire has 5 domains: mobility, self-care, usual activity, pain, and anxiety-depression. For each item, the subject selects one of 3 descriptive health states (from good to poor).
EuroQol-5 Dimensions index score | Up to 3 months
  European Quality of Life questionnaire consists of the EQ-5D index. The questionnaire has 5 domains: mobility, self-care, usual activity, pain, and anxiety-depression. For each item, the subject selects one of 3 descriptive health states (from good to poor).

SECONDARY OUTCOMES:
Functional capacity | Baseline
  The International Physical Activity Questionnaire (IPAQ) short form measures walking, moderate- and vigorous intensity, and total PA and daily time spent sitting on weekdays. PA was reported in MET·minutes/week and days per week and was scored using standardized IPAQ scoring protocols to yield total metabolic equivalent minutes (MET·minutes/week) of PA per week. Sitting time was reported as the amount of time in hours and/or minutes participants spent sitting on a weekday during the past seven days.
Functional capacity | Up to 7 days
  The International Physical Activity Questionnaire (IPAQ) short form measures walking, moderate- and vigorous intensity, and total PA and daily time spent sitting on weekdays. PA was reported in MET·minutes/week and days per week and was scored using standardized IPAQ scoring protocols to yield total metabolic equivalent minutes (MET·minutes/week) of PA per week. Sitting time was reported as the amount of time in hours and/or minutes participants spent sitting on a weekday during the past seven days.
Functional capacity | Up to 3 months
  The International Physical Activity Questionnaire (IPAQ) short form measures walking, moderate- and vigorous intensity, and total PA and daily time spent sitting on weekdays. PA was reported in MET·minutes/week and days per week and was scored using standardized IPAQ scoring protocols to yield total metabolic equivalent minutes (MET·minutes/week) of PA per week. Sitting time was reported as the amount of time in hours and/or minutes participants spent sitting on a weekday during the past seven days.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, Granada, Spain

IPD SHARING:
Plan to Share IPD: No